CLINICAL TRIAL: NCT07292896
Title: A Multicenter Study on the Normal Reference Range and Clinical Significance of the Right Atrioventricular Coupling Index Assessed by Artificial Intelligence-Based Three-Dimensional Echocardiography
Status: Not yet recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Other Study IDs: 3D-RACI-01
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy Adults; Pulmonary Hypertension; Tricuspid Regurgitation; Heart Failure; Atrial Septal Defect
Keywords: Right Atrioventricular Coupling Index; 3D Echocardiography; AI-assisted Imaging
MeSH Terms: conditions — Hypertension, Pulmonary; Tricuspid Valve Insufficiency; Heart Failure; Heart Septal Defects, Atrial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy Adults Group: Healthy adults aged 18 to 79 years are planned to be stratified into 6 age groups: 18-29 years, 30-39 years, 40-49 years, 50-59 years, 60-69 years, and ≥70 years. Each age group will include 120 participants of each sex.
- Pulmonary Hypertension Group: This group comprises adults with a confirmed diagnosis of mean pulmonary artery pressure (mPAP) ≥20 mmHg via right heart catheterization, in accordance with the diagnostic criteria for pulmonary hypertension specified in the 2022 ESC/ERS Guidelines.
- Tricuspid Regurgitation Group: Adults with moderate or severe primary/secondary tricuspid regurgitation confirmed by echocardiography.
- Atrial Septal Defect Group: Adults with atrial septal defect confirmed by echocardiography or transesophageal echocardiography, including non-intervened patients, those who underwent closure/surgical correction, and stable patients > 3 months after surgery.
- Heart Failure Group: Adults meeting the 2022 AHA/ACC/HFSA diagnostic criteria for heart failure are classified into three subgroups based on left ventricular ejection fraction (LVEF): heart failure with reduced ejection fraction (HFrEF, LVEF < 40%), heart failure with mildly reduced ejection fraction (HFmrEF, LVEF 40-49%), and heart failure with preserved ejection fraction (HFpEF, LVEF ≥ 50%).

SUMMARY:
This multicenter study aims to establish the normal reference range of the Right Atrioventricular Coupling Index (RACI) in healthy Chinese adults using AI-based 3DE technology. It will also analyze the correlation between RACI and physiological parameters such as age, gender, and body surface area. Additionally, the study will explore the variation characteristics of RACI in patients with pulmonary hypertension, heart failure, tricuspid regurgitation, and atrial septal defect, and evaluate the clinical value of RACI in disease diagnosis, differential diagnosis, and risk stratification.

ELIGIBILITY:
Healthy Adults Group

Inclusion Criteria:

* Participants must meet all of the following criteria to be enrolled:

  1. Of Han Chinese ethnicity
  2. Aged 18-79 years
  3. Normal blood pressure (< 140/90 mmHg)
  4. Normal fasting blood glucose
  5. Normal blood lipid levels (triglycerides, total cholesterol, low-density lipoprotein, high-density lipoprotein)
  6. Normal complete blood count results (hemoglobin concentration, white blood cell count, red blood cell count, platelet count)
  7. Normal liver and renal function (alanine transaminase < 2× upper limit of normal; normal creatinine and blood urea nitrogen)
  8. Normal electrocardiogram results (occasional atrial premature beats may be enrolled at the investigator's discretion)
  9. No structural heart disease and normal cardiac function confirmed by echocardiography

Exclusion Criteria:

Participants will be excluded if they meet any of the following criteria:

1. Clinically significant cardiac valve regurgitation (≥ mild severity)
2. Respiratory diseases: acute or chronic respiratory disorders
3. Endocrine diseases: thyroid disease, diabetes mellitus, hyperaldosteronism, pheochromocytoma, etc.
4. Abnormal liver function (alanine transaminase > 2× upper limit of normal), abnormal renal function (elevated creatinine beyond normal range), or dyslipidemia (elevated triglycerides, total cholesterol, low-density lipoprotein, or high-density lipoprotein)
5. Other systemic diseases: anemia, malignancy, connective tissue disease, large artery/peripheral vascular diseases (aortic dilation, aortic dissection, coarctation of the aorta, Takayasu arteritis, atherosclerosis), etc.
6. Pregnant or lactating women
7. Professional athletes
8. Poor-quality ultrasound images that cannot support parameter measurement and analysis

Pulmonary Hypertension Group

Inclusion Criteria:

Patients must meet all of the following criteria to be enrolled:

1. Aged 18-79 years
2. Confirmed diagnosis via right heart catheterization: mean pulmonary arterial pressure (mPAP) ≥ 20 mmHg, in accordance with the 2022 ESC/ERS guidelines

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria:

1. Unable to complete right heart catheterization or pressure-volume loop assessment
2. Complicated with significant left heart disease (left ventricular ejection fraction [LVEF] < 50%, significant mitral valve disease)
3. Pericardial disease or arrhythmias (e.g., atrial fibrillation) that severely impair right heart function evaluation
4. Poor-quality images that prevent accurate measurement of right atrial or right ventricular parameters
5. Concurrent liver or renal disease
6. Concurrent malignancy
7. History of surgical procedures such as pulmonary endarterectomy or balloon pulmonary angioplasty

Heart Failure Group

Inclusion Criteria:

Patients must meet all of the following criteria to be enrolled:

1. Aged 18-79 years
2. Meets the 2022 AHA/ACC/HFSA diagnostic criteria for heart failure

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria:

1.Complicated with significant valvular heart disease (e.g., severe mitral regurgitation, severe tricuspid regurgitation, etc.)

Tricuspid Regurgitation Group

Inclusion Criteria:

Patients must meet all of the following criteria to be enrolled:

1. Moderate or severe primary or secondary tricuspid regurgitation confirmed by echocardiography
2. Aged 18-79 years

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria:

1. Pericardial disease or arrhythmias (persistent atrial fibrillation) that interfere with measurements
2. Congenital heart disease or residual lesions after surgical correction

Atrial Septal Defect Group

Inclusion Criteria:

Patients must meet all of the following criteria to be enrolled:

1. Secundum atrial septal defect confirmed by echocardiography or transesophageal echocardiography
2. Patients who have not undergone closure or surgical correction, or stable patients with > 3 months postoperatively
3. Aged 18-79 years

Exclusion Criteria:

1.Complicated with other complex congenital heart diseases.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study enrolls 5 groups (18-79 years) from clinics/community:
  Healthy Adults: Han Chinese with normal cardiovascular function (vitals, labs, ECG, echo; no structural heart disease/systemic diseases/poor ultrasound).
  Pulmonary Hypertension: Diagnosed via right heart catheter (mPAP ≥20 mmHg, 2022 ESC/ERS); excluded if with left heart disease, interfering conditions, organ dysfunction, malignancy, or prior pulmonary surgery.
  Heart Failure: Meets 2022 AHA/ACC/HFSA criteria; excluded if with significant valvular disease.
  Tricuspid Regurgitation: Echo-confirmed moderate/severe regurgitation; excluded if with interfering pericardial/arrhythmic issues or congenital heart disease/residual lesions.
  Atrial Septal Defect: Echo/TEE-confirmed secundum defect (untreated or stable ≥3mo post-op); excluded if with complex congenital heart disease.
  All undergo standardized clinical/echo assessments for cardiac structure/function.
Sampling Method: Probability Sample
Enrollment: 2640 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Right Atrioventricular Coupling Index (RACI) | At study enrollment (baseline)
  RACI links the volumes of the right atrium (RA) and right ventricle (RV), with the degree of their volume matching reflecting their synergistic functional status during hemodynamic regulation

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Ma, MD, Principal Investigator — First Hospital of China Medical University
Locations (25):
- China (25):
  - Chongqing Liangjiang New Area Hospital of Traditional Chinese Medicine, Chongqing, Chongqing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - The Third Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang No.1 Peoples Hospital, Xiangyang, Hubei
  - The Second Affiliated Hospital of Jilin University, Changchun, Jilin
  - Anshan Central Hospital, Anshan, Liaoning
  - Ansteel Group General Hospita, Anshan, Liaoning
  - Chaoyang Central Hospital, Chaoyang, Liaoning
  - the Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Huludao Second People's Hospital, Huludao, Liaoning
  - Liaohua Hospital, Liaoyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Shaanxi University of Chinese Medicine, Xianyang, Shaanxi
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai

IPD SHARING:
Plan to Share IPD: No